CLINICAL TRIAL: NCT04575454
Title: Translational and Multimodal Brain Imaging of the Neural Correlates of Arousal and Awareness During Coma and Post-coma
Brief Title: Imaging of the Neural Correlates of Arousal and Awareness
Acronym: IMAGINA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_0672; 2020-A00375-34 (Other: IDRCB)
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-09

CONDITIONS: Lesional Coma
Keywords: coma; prognosis; diagnosis; functional imaging; PET-MRI; electrophysiology; eye-tracking
MeSH Terms: conditions — Coma; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comatose or post-comatose patients (Other)
  Interventions: Other: Multimodal evaluation of brain function : PET-MRI, electrophysiology, eye-tracking

INTERVENTIONS:
Other: Multimodal evaluation of brain function : PET-MRI, electrophysiology, eye-tracking — After 2 days of sedation withdrawal, each data should be collected within 3 days for organisation purposes :
  1. After installation and movement management with standardized routine care protocol: 18Fluoro-Desoxy-Glucose's infusion for PET
  2. Starting PET continuous acquisition
  3. Morphological MRI sequences
  4. MRI in Resting state N°1
  5. MRI DTI acquisition
  6. IRM in 2D-Arterial Spin Labelling
  7. IRM in Resting state 2
  8. End of PET continuous acquisition The day before or the day after PET-MR: standard 20 min EEG, somaesthetic evoked potentials, auditory evoked potentials, mismatch negativity, P300 oddball paradigm, local-global paradigm, P300 after music stimulation, EEG resting state for 10 min, CRS-R repeated before each examination (and at least 5 times for chronic patients), eye-tracking study of the environmental exploration.

SUMMARY:
In last decades, several advances in the neuro-intensive management have lead to decrease mortality in Intensive Care Units. A significant morbidity remains as patients survive after a traumatic coma with uncertain quality of awakening and a high risk of functional disability. Predicting awareness recovery and functional disability of those who will awake constitutes a major challenge to inform patients' relatives, to give the best chances in terms of rehabilitation resources or to adapt intensive cares to a reasonable level. Tools currently available are not sufficient neither to predict bad awakening outcome nor to predict good functional outcome. In many countries, life's support cessation is a constant call for robust evaluation as soon as possible in ICU but it is mandatory to reach a positive predictive value of non-awaking close to 100%. Many clinical, electro-physiological, biological, radiological and functional parameters have been conducted with comatose patients assuming the purpose to predict outcome. Regarding unfavourable outcome, the gold standard is the abolition of the N20 component of somatosensory evoked potentials but the specificity is high enough only for patients with anoxic coma. Several neurophysiological markers such as MMN, P300 are correlated to a favourable outcome but the sensitivity and specificity remains low for patients who suffered a severe traumatic brain injury. New Diffusion Tensor imaging sequences provide complementary information to detect small structural lesions (diffuse axonal lesions). Recently, functional MRI analyzing Resting State has also been proposed as a prognostic marker during coma. PET using Fluoro-Desoxy-Glucose is able to assess the metabolism in key regions of the awakening network in either anaesthesia or sleep. Recent studies have reported interesting results at the chronic stage but to our knowledge, these tools have only been used to address pathophysiology's issues and never to improve coma prognosis at the initial stage. We hypothesize that the heterogeneity of the population requires a global and accurate assessment of the central nervous system, combining structural, metabolic and functional information in order to refine the prognosis.

Our protocol integrates in one-sequence most radiological markers of brain injury within a unique PET-MRI in Lyon. Our most relevant originality consists in confronting FDG-PET and MRI sequences to a large clinical, electrophysiological and biological battery. The added clinical value would be to question the synergistic effect of each parameter and to find out which ones are the most useful for awakening prediction, as they have not been compared in a multi-parametric database.

PET-MRI, as a new device combining physiological and prognostic questioning, allows us:

* to implement a more integrative physio-pathological analysis
* to avoid the cofounding effect of awareness' fluctuations in recording simultaneously multiple functional imaging techniques.

The RS will be analyzed at 2 epochs in order to assess the stability of brain connectivity, related to neuronal activity (glucose metabolism) and brain perfusion.

The interest of imaging result will be compared across morphological and functional sequences and in comparison, to classical marker (clinical, electrophysiological and behavioural) to build the most precise prognostic tool for acute comatose patients in ICU or diagnostic/prognostic tool for chronic patients in rehabilitation unit.

ELIGIBILITY:
Inclusion Criteria:

Patients 1 Patients presenting either vascular or traumatic lesions or anoxic coma 2. For acute patients: Patients with no response to simple command 48h after sedation's cessation (coma, early vegetative state or MCS "minus") ; for chronic patients : patients without functional communication (including MCS "plus").

3. For acute patients: inclusion between 7 days (to reduce the effect of early oedema) and 30 days after the coma (to control the homogeneity of our cohort); for chronic patients: more than 3 months after anoxic coma or more than one year after 4. Patients included between 18 and 75 years old, to limit the risk of care withdrawal for poor previous medical condition 5. Patients evaluated by a global electrophysiological assessment at beside in ICU in a short delay before or after PET-MRI

Volunteers Healthy subjects:

1. Lack of neurological and / or psychiatric history, in particular without a history of head trauma with loss of consciousness lasting more than 30 min;
2. Participant between 18 and 75 years old matched in age and sex a posteriori with the patients
3. Subjects affiliated (or beneficiaries) to a social security scheme
4. Not subject to a legal protection measure;
5. Having given their free and informed consent to participate in the study in writing.
6. Subject having agreed to be registered in the national file of people who lend themselves to biomedical research

Exclusion Criteria:

Patients

1. Patient with an associated anoxic encephalopathy if the N20 response of SEP are not bilaterally abolished
2. Patients with contra-indication to MRI
3. Patients with hypersensibility to the active molecules (FDG) or to one of this excipient
4. Pregnant women
5. Minor patients
6. Patients under legal protection
7. Patients not affiliated to French health care system
8. Patients in poor medical condition (hemodynamic, respiratory instability)
9. Patients moribund or with previous decision of care withdrawal
10. Absence of relatives to give written consent

Volunteers Healthy subjects:

1. Subjects benefiting (or having benefited in the last month) from a medicinal treatment for somatic purposes having a cerebral or psychic impact (e.g. antihistamine); 2. Subjects with present or past dependence on alcohol or any other addictive substance according to DSM-IV-TR criteria, with the exception of nicotine and caffeine; 3.Subjects already participating in another biomedical research project or having participated for less than a year in a study using ionizing radiation; 4;Subjects with an inability to understand or carry out the study (language barrier, obvious lack of motivation, etc.) judged by the investigator 5.Minor patient; Patient under guardianship or curatorship; Patient not affiliated with French social security.

6.Pregnant woman or woman of childbearing age without proof of the absence of a current pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Awakening outcome at one year of coma onset | 12 months
  Predictive value of PET-MR multimodal assessment of brain function during early post-comatose period : Building a prognostic tool including miscellaneous parameters (clinical, biological, electrophysiological, metabolic PET and multimodal MRI) for the prediction of an unfavourable outcome (death, vegetative state, minimally conscious state) at 1 year post-coma.
  Describing the diagnostic utility of chronic disorder of consciousness classification and a late predictive value compared to the functional outcome at 1-year post-evaluation.

SECONDARY OUTCOMES:
Functional clinical evolution in presence of awareness (ordinal criteria within favorable outcome) defined by the Glasgow Outcome Scale - Extended (> 3, ranking from 4 - severe disability upper - to 8 - good recovery upper). | 12 months
  Building a prognostic tool including miscellaneous parameters (clinical, biological, electrophysiological, metabolic PET and multimodal MRI) for the prediction of cognitive and motor function when awakening appeared.

OTHER OUTCOMES:
Unfavorable clinical evolution in absence of awareness defined by the Glasgow Outcome Scale - Extended and further refined by the Coma Recovery Scale - Revised to distinguish Unresponsive Wakefulness Syndrome (UWS) from Minimally Conscious State (MCS) | 12 months
  Defining an association of criteria, which are available in the 1st month after coma, that are able to predict at 1 year with a high positive predictive value the level of disorder of consciousness in the subgroup with unfavourable outcome in analyzing (according to Coma Recovery Scale-Revised) the evolution of :
  * vegetative state patients
  * minimally-conscious patients
  * dead patients
Eye-tracking analysis of ocular exploration (combining pursuit and saccade eye movements) to assess cortical function based on temporal density (number of fixations per second) and topography (in an ecological visual field). | 12 months
  Defining the comparative diagnostic or prognostic value of clinical and eye-tracking based evaluation of the cortical function in acute and chronic phase of coma or post-coma, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: FLORENT GOBERT, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Hôpital Neurologique Pierre Wertheimer, Bron, France

IPD SHARING:
Plan to Share IPD: No